CLINICAL TRIAL: NCT05026125
Title: Quality Assessment of Orotracheal Intubation Without Neuromuscular Blocking Agents in Obese Patients with Two Doses of Remifentanil: a Pilot Study
Brief Title: Quality Assessment of Orotracheal Intubation Without Neuromuscular Blocking Agents in Obese Patients
Acronym: OBEREM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC31/20/0443; 2021-000727-12 (EudraCT Number)
Record Dates: First submitted 2021-08-23; First posted 2021-08-30 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Bariatric Surgery Candidate; Intubation Complication
Keywords: tracheal intubation; obese patient; neuromuscular blocking agent; remifentanil
MeSH Terms: conditions — Obesity | interventions — Remifentanil; Anesthesia; Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, double blinded and monocentric Pilot Study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: with randomization envelopes opened by the care provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group control (Active Comparator): 3 μg/kg (Ideal Body Weight) of Remifentanil
  Interventions: Drug: Remifentanil Injection
- Group Active (Experimental): 3 μg/kg (Ideal Body Weight) plus 30% of Remifentanil
  Interventions: Drug: Remifentanil Injection plus 30%

INTERVENTIONS:
Drug: Remifentanil Injection — Injection of 3 μg/kg (Ideal Body Weight) of Remifentanil in the induction phase of anesthesia for orotracheal intubation for bariatric surgery
  Other Names: orotracheal intubation; anesthesia; bariatric surgery
  Arms: Group control
Drug: Remifentanil Injection plus 30% — Injection of 3 μg/kg (Ideal Body Weight) plus 30% of Remifentanil in the induction phase of anesthesia for orotracheal intubation for bariatric surgery
  Other Names: orotracheal intubation; anesthesia; bariatric surgery
  Arms: Group Active

SUMMARY:
This study will assess the condition of orotracheal intubation in obese patients undergoing an elective bariatric surgery without the use of neuromuscular blocking agents.

During the induction of general anesthesia, Propofol - Remifentanil combination will be used.

The patients will be randomized in 2 groups with different doses of Remifentanil.

DETAILED DESCRIPTION:
The prevalence of obesity increases steadily. For anesthesiologists, the airway management of obese patients is known to be difficult and at risk. Tracheal intubation needs to be successful quickly. Neuromuscular blocking agents allow this option but with a risk of anaphylaxis and respiratory complications. In fact, for many surgical procedures those drugs are not necessary.

Numerous studies in non-obese patients with the combination of Remifentanil and Propofol have shown adequate conditions for tracheal intubation without neuromuscular blocking drugs. This combination has never been studied in obese patient.

After randomization, induction of general anesthesia will be performed with 2,5 mg/kg of Propofol in association with either 3 µg/kg of Ideal Body Weight of Remifentanil, or 3 µg/kg + 30% of Ideal Body Weight of Remifentanil.

Minutes after the induction, orotracheal intubation will be performed, and the Intubation Difficulty Scale recorded.

Other data on hemodynamic, respiratory and airway management will be are collected during the surgery.

In the Post Anaesthetic Care Unit (PACU),Any symptoms of traumatic airway management or aspiration are collected.

Those data will be again looked for and collected on the day of the patient's discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 and under 60 years old.
* ASA score ≤ 3
* Elective bariatric surgery for patient with BMI between 35 and 60 or elective revision of a bariatric surgery for patient with a BMI over 30.
* Patient with a written consent obtained with accurate information.

Exclusion Criteria:

* Patient with risk of aspiration
* Difficult airway known (Cormack score 3 ou 4).
* Opioids addiction.
* Alcoholism
* Chronic use of Opioids
* Confirmed Allergy to Propofol or Remifentanil
* Severe chronic hepatic, kidney or respiratory failure
* Patient already enrolled in another clinical study interfering with this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
percentage of patients with excellent conditions of intubation | Baseline
  Intubation conditions will be assessed using the intubation conditions score proposed by Viby-Mogensen and al. (Scandinavian score). The score defines intubation conditions: excellent (all variables are excellent), good (all variables are either excellent or good), or poor (presence of a poor variable).

SECONDARY OUTCOMES:
Hemodynamic effects : hypotension | Baseline
  Percentage of patients with arterial hypotension (>20% decrease in mean arterial pressure) within 40 minutes of intubation
Hemodynamic effects: bradycardia | Baseline
  Percentage of patients with bradycardia (>20% decrease in heart rate) within 40 minutes after intubation
Hemodynamic effects: use of vasopressor drugs | Baseline
  Number of times vasopressor drugs were used.after intubation
Respiratory effects: patients with desaturation day 0 | Baseline
  Percentage of patients with desaturation (pulse oximetry (SpO2) below 90%.)
Respiratory effects: patients with aspiration | From Baseline to day 2
  Percentage of patients with aspiration (defined by the existence of gastric fluid in the oropharynx during direct laryngoscopy or by the diagnosis of pneumopathy within 48 hours of surgery).
Intubation complexity | Baseline
  Intubation complexity Measured by Difficult intubation score (IDS): scale from 0 (easy) to >5 (very difficult)
Intubation difficulties with Cormack-Lehane classification | Baseline
  Intubation difficulties Measured by Cormack-Lehane classification (from 1: easy to 4 difficult)
Percentage of use of the study's emergency | Baseline
  Intubation difficulties measured by percentage of use of the study's emergency
Traumatic complications: anatomical lesion | Baseline
  Percentage of patients with an anatomical lesion (dental fracture, lip or mouth wound, oropharyngeal haemorrhage, vocal cord trauma)
Traumatic complications: postoperative functional discomfort | Day 2
  Percentage of patients with postoperative functional discomfort (laryngeal pain, aphonia or dysphonia).

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine FAURE, Md, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hospital University of Toulouse, Toulouse, France

REFERENCES:
- [Derived] Goudy P, Denis-Bonnin A, Thalamas C, Rousseau V, Migueres I, Faure G, Minville V. Quality of intubation using remifentanil in obese patients (OBEREM): a randomised, double-blind pilot trial. Anaesth Crit Care Pain Med. 2025 Nov 7:101673. doi: 10.1016/j.accpm.2025.101673. Online ahead of print. PMID 41207379